CLINICAL TRIAL: NCT06479720
Title: Efficacy and Safety of Solifenacin or Mirabegron With Local Estrogen Versus Combination Treatment With Mirabegron and Solifenacin for Refractory Overactive Bladder
Brief Title: Efficacy of Solifenacin or Mirabegron With Local Estrogen Versus Combination Pharmacotherapy for Overactive Bladder
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Mackay Memorial Hospital (Other)
Responsible Party: Principal Investigator, Hui-Hsuan Lau, MD, Head of urogynecology, Associate Professor, Mackay Memorial Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22MMHIS039e-3
Record Dates: First submitted 2024-06-23; First posted 2024-06-28 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2024-07

CONDITIONS: Effect of Drug; Urinary Bladder, Overactive
Keywords: Detrusor overactivity; Combined pharmacotherapy; Estrogens; Effectiveness
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Solifenacin Succinate; mirabegron; Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Solifenacin and mirabegron (Active Comparator): Solifenacin 5mg and Mirabegron 25mg
  Interventions: Drug: Combined pharmacotherapy with Solifenacin and Mirabegron
- Solifenacin with vaginal estrogen cream (Experimental): Solifenacin 5mg once per day with vaginal conjugated equine estrogen (CEE) 0.625 mg twice a week.
  Interventions: Drug: Solifenacin with vaginal estrogen cream
- Mirabegron with vaginal estrogen cream (Experimental): Mirabegron 25mg once per day with vaginal conjugated equine estrogen (CEE) 0.625 mg twice a week.
  Interventions: Drug: Mirabegron with vaginal estrogen cream

INTERVENTIONS:
Drug: Combined pharmacotherapy with Solifenacin and Mirabegron — Solifenacin (5mg) is anticholinergic and Mirabegron (25mg) is a beta-3 adrenergic agonist.
  Other Names: Vesicare and Betmiga
  Arms: Solifenacin and mirabegron
Drug: Solifenacin with vaginal estrogen cream — Solifenacin (5mg) is anticholinergic. Premarin, vaginal conjugated equine estrogen vaginal cream (0.625 mg).
  Other Names: Vesicare and Premarin
  Arms: Solifenacin with vaginal estrogen cream
Drug: Mirabegron with vaginal estrogen cream — Mirabegron (25mg) is a beta-3 adrenergic agonist. Premarin, vaginal conjugated equine estrogen vaginal cream (0.625 mg).
  Other Names: Betmiga and Premarin
  Arms: Mirabegron with vaginal estrogen cream

SUMMARY:
To investigates the effects of solifenacin or mirabegron with local estrogen versus combination treatment with solifenacin and mirabegron in women with overactive bladder

DETAILED DESCRIPTION:
Women with detrusor overactivity who were refractory to anti-muscarinics or mirabegron were enrolled for prospective study. Patients were divided into three groups: combined pharmacotherapy with solifenacin and mirabegron, solifenacin with vaginal estrogen cream and mirabegron with vaginal estrogen cream. Incontinence-related symptoms distress and impact on quality of life were evaluated by short form of Urinary Distress Inventory, (UDI-6), Incontinence Impact Questionnaire (IIQ-7) and Overactive Bladder Symptom Score (OABSS). Objective outcomes include changes from baseline in episodes of daily micturition, urgency, urinary incontinence and nocturia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with detrusor overactivity which defined as a urodynamic observation characterized by involuntary detrusor contractions during the filling phase. Those who were refractory to monotherapy with anti-muscarinics were enrolled for prospective study.

Exclusion Criteria:

* Postvoid urine retention before treatment
* Women who had medical illness and contraindication for using solifenacin and mirabegron, such as narrow-angle glaucoma and hypertension
* Concerns for using estrogen include: Women with history of cerebrovascular disease; thromboembolic disorders; gallbladder disease; known or suspected breast carcinoma; estrogen-dependent neoplasm or undiagnosed abnormal genital bleeding.

Ages: 40 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — The study focus on female overactive bladder.
Enrollment: 300 (Estimated)
Dates: Start 2022-06-16 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Short form of Urinary Distress Inventory (UDI-6) | Assess before treatment and 1 month, 3 months, 6 months and 1 year after treatment
  UDI-6 is a valid questionnaire, used particularly to investigate symptoms associated with lower urinary tract dysfunction and inquire on irritative, stress, and obstructive or discomfort complaints. UDI-6 consists of six items: frequent urination; leakage related to feeling of urgency; leakage related to activity, coughing, or sneezing; small amounts of leakage (drops); difficulty emptying the bladder; and pain or discomfort in the lower abdominal or genital area. The total score ranges from 0 to 18 , with a higher score indicating more severe of incontinence.
Short form of Incontinence Impact Questionnaire (IIQ-7) | Assess before treatment and 1 month, 3 months, 6 months and 1 year after treatment
  The IIQ-7 assess the impact of urinary incontinence on QoL. 7 items assess influence of urinary incontinence on physical activity, travel, social/relationships & emotional health. Each item is scored between 0 (activities not affected at all) to 3 (activities greatly affected). The total score ranges from 0 to 21, with a higher score indicating more severe of incontinence.
Overactive Bladder Symptom Score (OABSS) | Assess before treatment and 1 month, 3 months, 6 months and 1 year after treatment
  The total OABSS is the sum of four symptom scores: daytime frequency (score 0-2), nighttime frequency (score 0-3), urgency (score 0-5), and urgency incontinence (score 0-5). The total score ranges from 0 to 15, with a higher score indicating more severe of OAB symptoms.

SECONDARY OUTCOMES:
Episodes of daily micturition | Assess before treatment and 1 month, 3 months, 6 months and 1 year after treatment
  Patients report daily lower urinary tract symptoms episodes
Episodes of daily urgency | Assess before treatment and 1 month, 3 months, 6 months and 1 year after treatment
  Patients report daily lower urinary tract symptoms episodes
Episodes of daily incontinence | Assess before treatment and 1 month, 3 months, 6 months and 1 year after treatment
  Patients report daily lower urinary tract symptoms episodes
Episodes of daily nocturia | Assess before treatment and 1 month, 3 months, 6 months and 1 year after treatment
  Patients report daily lower urinary tract symptoms episodes

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Hsuan Lau, MD, Principal Investigator — Mackay Memorial Hospital
Locations (1):
- Mackay Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lightner DJ, Gomelsky A, Souter L, Vasavada SP. Diagnosis and Treatment of Overactive Bladder (Non-Neurogenic) in Adults: AUA/SUFU Guideline Amendment 2019. J Urol. 2019 Sep;202(3):558-563. doi: 10.1097/JU.0000000000000309. Epub 2019 Aug 8. PMID 31039103
- [Background] Mueller ER, van Maanen R, Chapple C, Abrams P, Herschorn S, Robinson D, Stoelzel M, Yoon SJ, Al-Shukri S, Rechberger T, Gratzke C. Long-term treatment of older patients with overactive bladder using a combination of mirabegron and solifenacin: a prespecified analysis from the randomized, phase III SYNERGY II study. Neurourol Urodyn. 2019 Feb;38(2):779-792. doi: 10.1002/nau.23919. Epub 2019 Jan 15. PMID 30644570
- [Background] Cardozo L, Lose G, McClish D, Versi E. A systematic review of the effects of estrogens for symptoms suggestive of overactive bladder. Acta Obstet Gynecol Scand. 2004 Oct;83(10):892-7. doi: 10.1111/j.0001-6349.2004.00581.x. PMID 15453881